CLINICAL TRIAL: NCT01291043
Title: Efficacy of Shiatsu in Pain, Flexibility, Sleep, Anxiety and Quality of Life in Individuals With Fibromyalgia: a Randomized Clinical Trial
Brief Title: Efficacy of Shiatsu in Individuals With Fibromyalgia: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Susan Yuan, MD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1297/09
Record Dates: First submitted 2011-01-27; First posted 2011-02-07 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Fibromyalgia
Keywords: Shiatsu; Fibromyalgia; Pain; Quality of sleep; Balance; Quality of life
MeSH Terms: conditions — Fibromyalgia; Pain; Sleep Initiation and Maintenance Disorders | interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shiatsu Group (Experimental)
  Interventions: Other: Shiatsu
- Control Group (No Intervention)

INTERVENTIONS:
Other: Shiatsu — 8-week treatment with two Shiatsu sessions per week (50-minute duration)
  Other Names: Acupressure
  Arms: Shiatsu Group

SUMMARY:
Fibromyalgia is a syndrome characterized by chronic and generalized musculoskeletal pain and tenderness in tender points. Its etiology and physiopathology are not well known; therefore its treatment is not satisfactory. Having this in view, a search for alternative and complementary medicine has been going on. This kind of practice is under pressure to present evidences of efficacy. A randomized clinical trial will be carried out with the aim of verifying the efficacy of a massage technique called Shiatsu in the improvement of pain, flexibility, quality of sleep, anxiety and quality of life of individuals with fibromyalgia. A sample of 34 subjects will be divided in Shiatsu Group and Control Group. All subjects will be evaluated in the beginning, in the middle and at the end of the treatment. Pain will be evaluated by the following instruments: visual analogue scale (VAS) and dolorimetry. The V-sit and reach test (VSRT) will be used to assess the flexibility of the hamstring muscles and lower back. The sleep will be evaluated with the Pittsburgh Sleep Quality Index (PSQI). The State-Trait Anxiety Inventory (STAI) will be used to evaluate anxiety. The evaluation of quality of life will be made with two instruments: fibromyalgia impact questionnaire (FIQ) and Activities-specific Balance Confidence (ABC) scale. In each treatment session, the subjects will be globally evaluated in the 14 main meridians and their respective points by touch, identifying points of excessive energy and their severity. The Control Group will wait for treatment and remain only with conventional pharmacological treatment, while the Shiatsu Group will receive a treatment with Shiatsu during eight weeks. The results will be expressed in mean and standard deviation. The normality of the data will be verified by the Shapiro-Wilk test. In the intragroup analysis, the T-test for the parametric data and the Wilcoxon test for the nonparametric data. In the comparison between groups, the analysis of variance (ANOVA) test will be used. The level of significance adopted will be α < 0.05.

DETAILED DESCRIPTION:
In the VAS, the subject marks the intensity of its pain in a 10 centimeter horizontal line.

In dolorimetry, the pain thresholds (PT) of 18 tender points are measured with the dolorimeter.

The VSRT assesses the flexibility mainly of the hamstring muscles and also of the lower back.

The PSQI is constituted of 19 questions. Scores of five or more indicate bad sleep quality and sleep disturbances.

The STAI is composed of two scales of items with semantic content which expresses the absence or presence of anxiety. Higher scores obtained in each scale indicate higher levels of anxiety.

The FIQ is composed of ten items. Higher scores indicate higher impact of fibromyalgia over quality of life The ABC scale was translated and adapted for this study and consists of a 17-item scale in which the level of confidence in balance is indicated in the execution of diverse activities.

ELIGIBILITY:
Inclusion Criteria:

* diagnoses of fibromyalgia

Exclusion Criteria:

* diagnoses of diseases that cause chronic pain
* skin lesions and infection
* pregnancy
* two consecutive absences in treatment sessions
* use of psychotherapy, physiotherapy or complementary therapies in the last 6 months
* regular supervised physical activity

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in VAS at 8 weeks | baseline and 8 weeks
  In the VAS the subject marks the intensity of its pain in a 10 centimeter horizontal line

SECONDARY OUTCOMES:
Change from baseline in FIQ at 4 weeks | baseline and 4 weeks
  The FIQ is composed of ten items, in which higher scores indicate higher impact of fibromyalgia over quality of life
Change from baseline in PSQI at 4 weeks | baseline and 4 weeks
  The sleep will be evaluated with the PSQI, which is constituted of 19 questions. Scores of five or more indicate bad sleep quality and sleep disturbances.
Change from baseline in STAI at 4 weeks | baseline and 4 weeks
  The STAI will be used to evaluate anxiety. It is composed of two scales of items with semantic content which expresses the absence or presence of anxiety. Higher scores indicate higher levels of anxiety.
Change from baseline in VSRT at 4 weeks | baseline and 4 weeks
  The VSRT will be used to assess the flexibility mainly of the hamstring muscles and also of the lower back.
Change from baseline in FIQ at 8 weeks | baseline and 8 weeks
  The FIQ is composed of ten items, in which higher scores indicate higher impact of fibromyalgia over quality of life.
Change from baseline in PSQI at 8 weeks | baseline and 8 weeks
  The sleep will be evaluated with the PSQI, which is constituted of 19 questions. Scores of five or more indicate bad sleep quality and sleep disturbances.
Change from baseline in STAI at 8 weeks | baseline and 8 weeks
  The STAI will be used to evaluate anxiety. It is composed of two scales of items with semantic content which expresses the absence or presence of anxiety. Higher scores indicate higher levels of anxiety.
Change from baseline in VSRT at 8 weeks | baseline and 8 weeks
  The VSRT will be used to assess the flexibility mainly of the hamstring muscles and also of the lower back.
Change from baseline in VAS at 4 weeks | Baseline and 4 weeks
  In the VAS, the subject marks the intensity of its pain in a 10 centimeter horizontal line.
Change from baseline in ABC scale at 4 weeks | baseline and 4 weeks
  The ABC scale was translated and adapted for this study and consists of a 17-item scale in which the level of confidence in balance is indicated in the execution of diverse activities.
Change from baseline in ABC scale at 8 weeks | baseline and 8 weeks
  The ABC scale was translated and adapted for this study and consists of a 17-item scale in which the level of confidence in balance is indicated in the execution of diverse activities.
Change from baseline in PT mean at 4 weeks | baseline and 4 weeks
  In dolorimetry, the PT of 18 tender points are measured with the dolorimeter. Then the PT mean will be calculated.
Change from baseline in PT mean at 8 weeks | baseline and 8 weeks
  In dolorimetry, the PT of 18 tender points are measured with the dolorimeter. Then the PT mean will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Susan LK Yuan, MSc, Principal Investigator — Faculty of Medicine of the University of Sao Paulo; Amelia P Marques, PhD, Study Director — Faculty of Medicine of the University of Sao Paulo
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil